CLINICAL TRIAL: NCT02847702
Title: A Phase 2a, Multicenter, Randomized, Double-blind, Placebo Controlled and Active-controlled, Parallel-group Study Evaluating the Analgesic Efficacy and Safety of VM902A in Subjects With Moderate to Severe Chronic Pain Due to Osteoarthritis of the Knee
Brief Title: A Study to Evaluate the Analgesic Efficacy and Safety of VM902A in Subjects With Osteoarthritis (OA) of the Knee
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TKA2001
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Osteoarthritis Pain of the Knee
Keywords: Osteoarthritis; Pain; Osteoarthritis, knee
MeSH Terms: conditions — Osteoarthritis; Pain; Osteoarthritis, Knee | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- VM902A 200 mg (Experimental): VM902A 200-mg Capsules
  Interventions: Drug: VM902A 200-mg Capsules; Drug: Placebo
- VM902A 400 mg (Experimental): VM902A 400-mg Capsules (2 x 200-mg capsules)
  Interventions: Drug: VM902A 400-mg Capsules; Drug: Placebo
- Naproxen (Active Comparator): Naproxen 500-mg Capsules
  Interventions: Drug: Naproxen 500-mg Capsules; Drug: Placebo
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VM902A 200-mg Capsules — Taken orally with food twice daily
  Arms: VM902A 200 mg
Drug: VM902A 400-mg Capsules — Taken orally with food twice daily
  Arms: VM902A 400 mg
Drug: Naproxen 500-mg Capsules — Taken orally with food twice daily
  Arms: Naproxen
Drug: Placebo — Capsules to match VM902A and/or naproxen taken orally with food twice daily

SUMMARY:
The purpose of this study is to evaluate the analgesic efficacy, safety, and tolerability of VM902A twice daily compared to placebo in subjects with moderate to severe chronic pain due to OA of the knee.

ELIGIBILITY:
Key Inclusion Criteria Include:

1. Males and females ≥ 40 and ≤ 75 years of age with moderate to severe chronic OA pain of the knee (lasting several hours daily) as their predominant pain condition for at least 6 months prior to screening
2. Diagnostic criteria for primary pain condition (American College of Rheumatology [ACR] clinical and radiographic criteria):

   * At least 1 of the following in addition to knee pain: age > 50, stiffness < 30 min, crepitus on active motion, and
   * Kellgren-Lawrence (K-L) grade 2 or 3 radiographic evidence at the screening visit as determined by a local radiologist or rheumatologist. Note that K-L grades 2 to 3 require the presence of osteophytes, which is required to meet ACR clinical and radiographic criteria for knee OA
3. Subjects whose OA pain of the index knee is not adequately treated prior to the screening visit:

   • Subjects must have a self-reported average pain intensity rating of moderate or severe on a verbal rating scale (ie, none, mild, moderate, and severe) over the 7 days prior to the screening visit
4. The subjects must have "average pain over the last 24 hours" scores ≥ 5 and ≤ 9 on an 11-point numerical rating scale (NRS) for the index knee on ≥ 3 consecutive days during the screening period and come in for randomization within 72 hours after qualification is met
5. Subjects who are willing and able to stop taking any/all analgesic medications, including over-the-counter pain medications, opioids, marijuana, and topical analgesics for OA pain for the duration of the treatment period, with the exception of study-specific rescue medication.

Key Exclusion Criteria Include:

1. Subjects with radiographic evidence of OA with K-L grade 0, 1, or 4
2. Subjects at risk for destructive arthropathy, subjects with a history of osteonecrosis, osteoporotic fracture, rapidly progressive osteoarthritis (RPOA 1 and 2), subchondral insufficiency fracture, and hip/knee dislocations
3. Subjects considered high risk for surgery based upon American Society of Anesthesiologists physical classification system for surgery grading, or subjects who would not be willing to undergo joint replacement surgery if required
4. Subjects with chronic pain conditions other than OA of the knee as their predominant pain condition, including gout (except for subjects with gout that is controlled with diet and/or with stable suppressive treatment with uric acid reducing medication(s) and/or colchicine, and who have not had any attack within the past 2 years), pseudogout, psoriatic arthritis, active Lyme disease, rheumatoid arthritis or any other inflammatory arthritis, fibromyalgia, neuropathic pain conditions, bursitis, or acute injury or signs of active infection in the target pain area
5. Subjects scheduled for surgical interventions of the disease site or any other major surgery during the study conduct period
6. Subjects with a history of a prior joint replacement of the index knee
7. Subjects who have had arthroscopy on either knee or hip within 6 months of entering the study, or open surgery on either knee or hip within 12 months of entering the study.

Other protocol-specific inclusion/exclusion criteria may apply.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-11-22 (Actual); Study Completion 2016-11-22 (Actual)

PRIMARY OUTCOMES:
Daily "Average Pain Over the Last 24 Hours" Score at Week 4 | Week 4

SECONDARY OUTCOMES:
Weekly "Average Pain Over the Last 24 Hours" at Week 4 | Week 4
Average Daily "Pain Right Now" Score at Week 4 | Week 4
Western Ontario and McMaster OA Index (WOMAC) - Total Scores | Week 4
Western Ontario and McMaster OA Index (WOMAC) Pain Severity Subscale Score | Week 4
Western Ontario and McMaster OA Index (WOMAC) Physical Function Subscale Score | Week 4
Western Ontario and McMaster OA Index (WOMAC) Stiffness Subscale Score | Week 4
Modified Brief Pain Inventory-Short Form (mBPI-SF) - Total Scores | Week 4
Modified Brief Pain Inventory-Short Form (mBPI-SF) Pain Severity Subscale Score | Week 4
Modified Brief Pain Inventory-Short Form (mBPI-SF) Pain Interference Subscale Score | Week 4
Medical Outcomes Study 36-item Short-Form Health Survey (SF-36) | Week 4
EuroQol-5D (EQ-5D) to Measure Health Status | Week 4
Patient Global Impression of Change (PGIC) at the End of the Double-blind Period | Week 4
Supplemental Analgesic Medication Use | Days 1 - 28
  The average daily number of tablets of supplemental pain medication taken during the study.
Responder to Treatment | Week 4
  The percentage reduction from the baseline mean "average pain over the last 24 hours" score to the week 4 mean pain score from the mBPI-SF pain severity subscale.
Hospital Anxiety and Depression Scale (HADS) Score | Baseline to Week 4
  Safety assessment to evaluate the impact of VM902A on mood (anxiety and depression)
Columbia-Suicide Severity Rating Score (C-SSRS) | Baseline to Week 4
  Safety assessment to evaluate the occurrence of treatment-emergent suicidal ideation
Survey of Autonomic Symptoms (SAS) Score | Baseline to Week 4
  Safety assessment to evaluate symptoms of autonomic dysfunction
Kellgren-Lawrence Classification (K-L) Score | Baseline to Week 4
  Safety assessment to classify the severity of knee OA

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Investigational Site, Birmingham, Alabama
  - Investigational Site, Huntsville, Alabama
  - Investigational Site, DeLand, Florida
  - Investigational Site, Hialeah, Florida
  - Investigational Site, Homestead, Florida
  - Investigational Site, Jupiter, Florida
  - Investigational Site, Orlando, Florida
  - Investigational Site, Port Orange, Florida
  - Investigational Site, Port Saint Lucie, Florida
  - Investigational Site, The Villages, Florida
  - Investigational Site, West Palm Beach, Florida
  - Investigational Site, Columbus, Georgia
  - Investigational Site, Avon, Indiana
  - Investigational Site, Muncie, Indiana
  - Investigational Site, Newton, Kansas
  - Investigational Site, Prairie Village, Kansas
  - Investigational Site, New Bedford, Massachusetts
  - Investigational Site, Bay City, Michigan
  - Investigational Site, Troy, Michigan
  - Investigational Site, Kansas City, Missouri
  - Investigational Site, St Louis, Missouri
  - Investigational Site, Hartsdale, New York
  - Investigational Site, Rosedale, New York
  - Investigational Site, The Bronx, New York
  - Investigational Site, Cincinnati, Ohio
  - Investigational Site, Dayton, Ohio
  - Investigational Site, Dublin, Ohio
  - Investigational Site, Duncansville, Pennsylvania
  - Investigational Site, Ogden, Utah
  - Investigational Site, Salt Lake City, Utah
  - Investigational Site, South Jordan, Utah

IPD SHARING:
Plan to Share IPD: No